CLINICAL TRIAL: NCT06771336
Title: Standard of Care Pathways Evaluation of Patients Treated for Facial Reconstruction After Surgery for Head and Neck Cancer, Using the Conventional Technique (Free Bone Flap): a Medico-economic Study
Brief Title: Biomedical Innovation for Facial Bone Reconstruction in Oncology: BIOFACE PASS a Medico-economic Study Describing the Standard Pathway of Patients Treated by Free Bone Flap
Acronym: BIOFACE PASS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0307; 2024-A01597-40 (Other: Agence National de Sécurité du Médicament)
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancers
Keywords: Mandibullar or maxillar reconstruction; Care pathway; Free bone flap; Medico-economic study
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with oral cavity cancer or maxillary and/or oropharynx cancer: Patients with oral cavity cancer or maxillary and/or oropharynx cancer eligible for treatment by surgery requiring a mandibulectomy or segmental maxillectomy and having a free bone flap for facial reconstruction.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Quality of life questionnaires, questionnaires for assessing functional results, micro-costing questionnaire, informal support assessment questionnaires

SUMMARY:
The purpose of this study is to describe the standard of care pathway of patients treated by free bone flap for facial mandibullar or maxillar reconstruction after surgery for head and neck cancers.

DETAILED DESCRIPTION:
Curative management of head and neck cancers frequently requires an interrupting mandibulectomy or maxillectomy. Surgery may involve resection of anatomical structures such as jaw or maxilla. The use of free vascularized fibula or scapula flap is the "gold standard" for mandibular and maxillary reconstruction but remains suboptimal as resulting in difficulty in speaking, swallowing, and disfigurement.

The BIOFACE project, funded by "Appel à Projet -Recherche Hospitalo-Universitaire en santé (RHU)" number 6 France 2023, aims to develop a new biomaterials based device to reconstruct these structure after surgery. In addition to the clinical benefits, this project aims to demonstrate the medico-economic benefits of the BIOFACE solution. Therefore, the Bioface PASS study has been designed to describe standard of care pathways of patients treated by free bone flap for facial reconstruction after surgery for head and neck cancer. Direct medical and non-medical costs, and daily allowance 12 months after the end of treatment, and quality of life will be recorded at the inclusion, 3 and 12 months.

From the hospital perspectives, production costs will be recorded using the micro-costing approach.

ELIGIBILITY:
Inclusion Criteria:

* Patient with oral cavity cancer or maxillary and/or oropharynx cancer
* Eligible for treatment by surgery requiring a mandibulectomy or segmental maxillectomy and having a free bone flap for facial reconstruction.
* Patient whose disease is classified Stage cT4a, N0 to N3, M0
* Treatment with a feasible curative aim (no contraindication to optimal treatment such as surgery or chemotherapy at a curative dose)
* Age greater than or equal to 18 years
* Patient affiliated to a Social Security scheme in France
* Patient having given written informed consent

Non-inclusion Criteria:

* Patient having any situation considered by the doctor as a reason for non-inclusion such as stenosis of the leg tripod not allowing reconstruction by fibula, one or more comorbidity(s) not allowing reconstruction by free bone flap or making this reconstruction too much risk
* Patient having had previous radiotherapy
* Patient with severe coagulation disorders
* Patients deprived of liberty or under legal protection regime (curatorship and guardianship, safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participation in the protocol will be offered to all patients meeting the eligibility criteria during the 3-year inclusion period.
  It is planned to include 200 operated patients, including 50 treated by maxillectomy and 150 treated by mandibulectomy.
  Nine French cancer centers and university hospitals will participate in the project: the University Hospitals of Toulouse, Amiens, Rouen, Lille, Montpellier, Nantes, the Gustave Roussy Institute, the Antoine Lacassagne Center (Nice) and the Hospices Civil de Lyon.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Description of the standard of care pathway of patients treated by free bone flap for facial mandibullar or maxillar reconstruction after surgery for head and neck cancers | 12 months
  The primary outcome measure is a composite endpoint consisting of the description of care pathways based on care consumption (scheduled and unscheduled hospitalizations and consultations, medical procedures and medications).
  The study of pathways will take into account data from the National Health Data System (i.e. healthcare consumption).
  These data will then be aggregated and structured to form time sequences representing the care pathways (and classes of care pathways) of patients using the optimal matching method. These sequences will include several medical events such as consultations, treatments, hospitalizations for example. This will provide us with a simplified but detailed representation of care trajectories. The individual care sequences thus constructed will allow us to carry out sequence analyzes aimed at creating patient clusters.

CONTACTS AND LOCATIONS:
Overall Officials: Agnès DUPRET-BORIES, Principal Investigator — University Hospital, Toulouse
Locations (9):
- France (9):
  - University hospital of Amiens- Picardie, Amiens
  - University hospital of Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - University hospital of Montpellier, Montpellier
  - University hospital of Nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - University hospital of Rouen, Rouen
  - University hospital of Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif